CLINICAL TRIAL: NCT06913699
Title: The Ameliorative Effect of C-Kit (+) Hepatic Endothelial Cells With Mertk Deficiency on Nonalcoholic Steatohepatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: Approval No.2024YS-050
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Liver biopsy tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Ultrasonund-guided percutaneous liver biopsy — All patients completed blood routine, coagulation function and liver biochemical indexes before surgery, and informed the patients and their families about the purpose and risks of surgery, and signed an informed consent. During the procedure, the patient was placed in the left lateral decubitus position. After locating by ultrasound and routine disinfection, 0.5% lidocaine was used for local anesthesia. Under the guidance of ultrasound, a 16G disposable biopsy needle (SC1620) was inserted into the liver parenchyma, and the biopsy gun was started and fired for sampling. The removed liver tissue was fixed in 4% formaldehyde solution and sent to the pathology department. The patient's puncture site was disinfected and covered with sterile dressing, and the abdominal band was bandaged. The patients were instructed to stay in bed for 24 hours after operation, closely observe whether there was pain and bleeding after operation, and monitor electrocardiogram for 24 hours.

SUMMARY:
The prevalence of non-alcoholic fatty liver disease (NAFLD) has been steadily increasing, with 10-20% of affected individuals progressing to non-alcoholic steatohepatitis (NASH). NASH is pathologically characterized by hepatic inflammation, steatosis, and hepatocyte injury. Furthermore, this condition carries a significant risk of progression to advanced hepatic fibrosis (pathological Scheuer fibrosis stage F≥3), cirrhosis, and even hepatocellular carcinoma (HCC). In recent years, NASH has emerged as the leading contributor to the growing burden of cirrhosis worldwide, representing a major public health challenge. Despite the high incidence and clinical severity of NAFLD, there are currently no FDA-approved therapeutic agents for its management. Therefore, elucidating the molecular mechanisms underlying NAFLD-associated NASH progression is critical for developing targeted pharmacological interventions capable of preventing, ameliorating, or potentially reversing disease progression.

DETAILED DESCRIPTION:
I. Study Background Non-alcoholic fatty liver disease (NAFLD) has become one of the most prevalent liver disorders globally. Despite its high incidence and severity, no effective therapeutic agents currently exist. Existing treatments focus on symptomatic relief, such as hepatoprotection and enzyme reduction, rather than addressing the underlying pathogenesis. Therefore, elucidating the mechanisms driving the progression of NAFLD-related non-alcoholic steatohepatitis (NASH) and hepatic fibrosis is critical for developing preventive, ameliorative, or even curative strategies, holding significant strategic importance.

1. Role of LSECs in NAFLD Pathogenesis:

   Liver sinusoidal endothelial cells (LSECs), the primary components of the hepatic sinusoidal endothelium, form a physical barrier regulating substance exchange between the hepatic parenchyma and circulation. As highly specialized endothelial cells (ECs) and the most abundant non-parenchymal cells (NPCs) in the liver, LSECs play pivotal roles in hepatic pathophysiology. Targeting LSEC function represents a promising approach to mitigate NAFLD progression and complications.
2. Heterogeneous Transcriptomic Features of LSEC Subpopulations in NAFLD:

   Single-cell RNA sequencing (scRNA-seq) enables genome-wide amplification and sequencing at the single-cell level. In the liver, hepatocytes (HCs) and NPCs exhibit marked transcriptomic heterogeneity, underpinning metabolic and functional zonation. This highlights the potential of single-cell analysis in understanding liver diseases. However, scRNA-seq studies on LSECs in NAFLD remain unexplored.
3. Hypothesis: C-Kit(+)/Gas6(-)-LSEC Subpopulation Exacerbates NAFLD via Gas6/Mertk-Mediated Regulation of PINK1 Mitophagy:

Bone marrow-derived endothelial progenitor cells (EPCs), marked by C-Kit (CD117), may express C-Kit in ECs under pathological conditions. Gas6, a ligand for TAM receptors (Tyro3, Axl, Mertk), activates downstream signaling cascades regulating cell migration, inflammation, survival, and mitophagy. In NAFLD, Gas6/Mertk exhibits cell-specific roles : Anti-inflammatory in hepatic macrophages; Pro-fibrotic in hepatic stellate cells (HSCs); Protective in hepatocytes (HCs). However, the role of Gas6/Mertk in LSECs during NAFLD remains unknown. Mitochondrial dysfunction is a hallmark of NAFLD, and impaired mitophagy (e.g., PINK1 deficiency) exacerbates hepatic inflammation, steatosis, and fibrosis. Emerging evidence suggests Gas6/Mertk enhances mitophagy to preserve mitochondrial function. For instance, Mertk-/- mice exhibit cardiomyocyte mitochondrial dysfunction, and Gas6 promotes mitophagy.

Our preliminary scRNA-seq data from HFD/ND mice identified a unique C-Kit(+)/Gas6(-)-LSEC subpopulation. These LSECs induced mitophagy impairment in co-cultured HCs/HSCs, manifesting as mitochondrial senescence, oxidative stress, HSC activation, HC lipid deposition, and inflammation. Investigating how this subpopulation drives NAFLD progression will unveil novel pathophysiological mechanisms and therapeutic targets, forming the basis of this study.

II. Study Objectives To elucidate the expression levels of C-Kit and Gas6/Mertk ligand-receptor pairs in liver tissues of NAFLD patients.

III. Study Procedures

(1) Inclusion and Exclusion Criteria

1. Inclusion Criteria: NAFLD diagnosis per Guidelines for the Prevention and Treatment of Non-Alcoholic Fatty Liver Disease (2018 Edition). Age 18-65 years.
2. Exclusion Criteria: Cirrhosis (compensated or decompensated), hepatocellular carcinoma, active viral hepatitis (HBV, HCV), primary biliary cholangitis, primary sclerosing cholangitis, recent history of illicit drug use, alcohol intake≥20 g/day for women and ≥30 g/day for men, current pregnancy or breastfeeding, severe comorbidities.

(2) Study Design

1. Liver Biopsy and Tissue Collection:

   Ultrasound-guided liver biopsy in 6 NAFLD patients. Histopathological evaluation (HE, Masson staining) for NASH and fibrosis (NAS and Scheuer scoring). Clinical data collection and liver tissue storage (-80°C).
2. Expression Analysis of C-Kit and Mertk:

Immunofluorescence co-staining of liver tissues. 3. Statistical Analysis: Compare C-Kit and Mertk expression levels in mild and severe NAFLD patients.

(3) Enrollment and Workflow

1. Baseline Data Collection:

   ①Demographic and clinical parameters: name, sex, age, ethnicity, birthdate, height, weight, disease onset, contact information.

   ② Laboratory tests: CBC, ALT, AST, TBIL, TG, cholesterol, glucose, total protein, albumin.

   ③Clinical assessments: blood pressure, BMI, abdominal ultrasound, FibroScan.
2. Biopsy Protocol:

   * Ultrasound-guided percutaneous liver biopsy within 1 month of enrollment. ②Tissue specimen requirements: ≥3 mm diameter, 5-8 mm length. ③Storage: -80°C for C-Kit and Mertk gene analysis.

IV. Expected Outcomes Clarify the regulatory relationship between C-Kit (+) LSECs and the Gas6-Mertk signaling pathway in NAFLD patient liver tissues.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Non-Alcoholic Fatty Liver Disease
* Age 18-65 years

Exclusion Criteria:

* Cirrhosis (compensated or decompensated)
* Hepatocellular carcinoma
* Active viral hepatitis (HBV, HCV)
* Primary biliary cholangitis
* Primary sclerosing cholangitis
* Recent history of illicit drug use
* Alcohol intake≥20 g/day for women and ≥30 g/day for men
* Current pregnancy or breastfeeding
* Severe comorbidities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised adults with NAFLD confirmed by imaging (ultrasound, CT, or MRI), excluding secondary causes (e.g., alcohol consumption >30/20 g/day for men/women, viral hepatitis, or steatogenic medications). . Exclusion criteria included Cirrhosis (compensated or decompensated), hepatocellular carcinoma, primary biliary cholangitis, primary sclerosing cholangitis, recent history of illicit drug use, current pregnancy or breastfeeding, severe comorbidities. NAFLD severity was categorized using non-invasive fibrosis scores (NFS) or liver biopsy (steatosis, inflammation, fibrosis staging).
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mertk expression levels of liver tissues | From enrollment to the end of treatment at 4 weeks
  1. Liver Biopsy and Tissue Collection:
     Ultrasound-guided liver biopsy in 6 NAFLD patients. Histopathological evaluation (HE, Masson staining) for NASH and fibrosis (NAS and Scheuer scoring). Clinical data collection and liver tissue storage (-80°C).
  2. Expression Analysis of Mertk:
     Immunofluorescence staining of liver tissues.
  3. Statistical Analysis:
  Compare Mertk expression levels between mild and severe NAFLD patients.
C-Kit expression levels of liver tissues | From enrollment to the end of treatment at 4 weeks
  1. Liver Biopsy and Tissue Collection:
     Ultrasound-guided liver biopsy in 6 NAFLD patients. Histopathological evaluation (HE, Masson staining) for NASH and fibrosis (NAS and Scheuer scoring). Clinical data collection and liver tissue storage (-80°C).
  2. Expression Analysis of C-Kit:
     Immunofluorescence staining of liver tissues.
  3. Statistical Analysis:
  Compare C-Kit expression levels between mild and severe NAFLD patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital (East Hospital Affiliated To Tongji University), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes